CLINICAL TRIAL: NCT03721367
Title: Prospective Cross-Sectional Non-invasive Assessment of Chronic Liver Disease in Urea Cycle Disorders
Brief Title: Chronic Liver Disease in Urea Cycle Disorders
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Seattle Children's Hospital (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Lindsay Burrage, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-40988; UCDC 5118 (Other: Urea Cycle Disorders Consortium)
Record Dates: First submitted 2018-06-20; First posted 2018-10-26 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Urea Cycle Disorder
MeSH Terms: conditions — Urea Cycle Disorders, Inborn | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urea Cycle Disorders
  Interventions: Other: Diagnostic Ultrasound

INTERVENTIONS:
Other: Diagnostic Ultrasound — All individuals will undergo a blood draw for measurement of biomarkers of liver disease and an ultrasound with shear-wave elastography.

SUMMARY:
This is a pilot, cross-sectional study to assess liver stiffness and markers of hepatic injury, function, and fibrosis in patients with urea cycle disorders. This study will be conducted at 3 UCDC sites: Baylor College of Medicine in Houston, Texas, University of California San Francisco (UCSF), San Francisco, California and Seattle Children's Hospital, Seattle,Washington

DETAILED DESCRIPTION:
Urea cycle disorders (UCDs) are among the most common inborn errors of liver metabolism.With early diagnosis and improved treatments, the survival of individuals with UCDs has improved, and this improved survival has led to unmasking of some long-term complications such as hepatic dysfunction and progressive fibrosis in a subset of patients. Hepatic complications in UCDs are quite variable and dependent upon the specific metabolic defect. Currently, there are no guidelines for monitoring hepatic complications or extent of liver disease in UCDs.

The purpose of this study is: 1) To determine whether liver stiffness is higher in individuals with ASS1D, ASLD, and ARG1D as compared to females with OTCD, and to assess liver stiffness in other UCDs (citrin deficiency, NAGSD, CPS1D, and males with OTCD), 2) To test whether markers of hepatocellular injury and function and novel serum biomarker panels for hepatic fibrosis provide evidence of chronic liver disease in individuals with ASS1D, ASLD, and ARG1D as compared to OTCD and to assess these sample markers of hepatocellular injury and function and novel serum biomarker panels for hepatic fibrosis in other UCDs (citrin deficiency, NAGSD, CPS1D, and males with OTCD).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 5 years and < 60 years
2. Weight ≥ 11 kg
3. Males or females with a diagnosis of OTCD based on molecular or enzymatic testing. Males or females with a diagnosis of CPS1D, citrin deficiency, NAGSD, ASS1D, ASLD or ARG1D based on biochemical OR molecular, OR enzymatic testing

Exclusion Criteria:

1. History of hyperammonemia (blood ammonia greater than 100 micromoles/L) documented in the medical record or reported by the patient in the 30 days preceding enrollment visit
2. History of Liver transplantation
3. Current pregnancy
4. Confirmed diagnosis of chronic viral hepatitis, autoimmune liver disease, or alcohol liver disease

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with urea cycle disorders
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagamani SCS, Ali S, Izem R, Schady D, Masand P, Shneider BL, Leung DH, Burrage LC. Biomarkers for liver disease in urea cycle disorders. Mol Genet Metab. 2021 Jun;133(2):148-156. doi: 10.1016/j.ymgme.2021.04.001. Epub 2021 Apr 8. PMID 33846069
- [Derived] Burrage LC, Madan S, Li X, Ali S, Mohammad M, Stroup BM, Jiang MM, Cela R, Bertin T, Jin Z, Dai J, Guffey D, Finegold M; Members of the Urea Cycle Disorders Consortium (UCDC); Nagamani S, Minard CG, Marini J, Masand P, Schady D, Shneider BL, Leung DH, Bali D, Lee B. Chronic liver disease and impaired hepatic glycogen metabolism in argininosuccinate lyase deficiency. JCI Insight. 2020 Feb 27;5(4):e132342. doi: 10.1172/jci.insight.132342. PMID 31990680

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Urea Cycle Disorders
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Urea Cycle Disorders
Number analyzed (Participants) | 28
Age, Continuous [Mean (Full Range); unit: years] | 15 [5 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13
  Native American | 2
  Hispanic | 9
  African-American | 3
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 28
UCD diagnosis [Count of Participants; unit: Participants]
  OTC Deficiency (Male) | 3
  OTC Deficiency (Female) | 7
  ASS1 Deficiency | 4
  ASL Deficiency | 8
  ARG1 Deficiency | 6
BMI [Count of Participants; unit: Participants]
  Underweight | 1
  Healthy | 12
  Overweight | 5
  Obese | 10
History of Hyperammonemia [Count of Participants; unit: Participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: Liver Stiffness as Measured by Shear Wave Elastography
Description: Shear wave elastography in m/s is a measure of liver stiffness, a surrogate measure for hepatic fibrosis. Normal liverstiffness is < 1.35 m/s and abnormal liver stiffness is >1.35 m/s
Time Frame: One measurement made on the day of study visit
Population: The data for this outcome was reliable for only 27 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Urea Cycle Disorders
Number analyzed (Participants) | 27
Participants
  Normal Liver Stiffness | 13
  Abnormal Liver Stiffness | 14

2. Primary Outcome: Grey Scale Ultrasound Findings
Description: Grey scale ultrasound findings
Time Frame: Baseline, once
Measure: Count of Participants; unit: Participants
Arm/Group | Urea Cycle Disorders
Number analyzed (Participants) | 28
Participants
  Normal hepatic parenchyma on grey scale ultrasound | 15
  Abnormal hepatic parenchyma on grey scale ultrasound | 13

3. Secondary Outcome: Fibrotest
Description: Fibrotest is a blood test that is a surrogate measure for hepatic fibrosis. F0 is normal. >F0 predicts at least minimal fibrosis.
Time Frame: Baseline, once
Measure: Count of Participants; unit: Participants
Arm/Group | Urea Cycle Disorders
Number analyzed (Participants) | 28
Participants
  F0 | 19
  >F0 | 9

ADVERSE EVENTS:
Time Frame: Baseline study visit
Arm/Group | Urea Cycle Disorders
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03721367/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT03721367/SAP_001.pdf